CLINICAL TRIAL: NCT01847768
Title: Comparison of Airway Remodeling Mediators Following Experimental Human Rhinovirus Infection in Subjects With Mild to Moderate Asthma, and in Healthy, Non-asthmatic Control Subjects (AADCRC-UC-01)
Brief Title: Human Rhinovirus Infection and Airway Remodeling Mediators
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Asthma and Allergic Diseases Cooperative Research Centers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DAIT AADCRC-UC-01; AADCRC-UC-01 (Other: Asthma and Allergic Diseases Cooperative Research Centers)
Record Dates: First submitted 2013-05-01; First posted 2013-05-07 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
Keywords: asthma; rhinovirus; remodeling mediators; human rhinovirus infection
MeSH Terms: conditions — Asthma | interventions — viral protein 1, rhinovirus; Cold Temperature; Bronchoalveolar Lavage; Nasal Lavage; Phlebotomy; Blood Specimen Collection; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthmatic Group (Experimental): Subjects with well-controlled, mild-moderate allergic asthma.Subjects will be inoculated with a total dose of 1000 TCID50 of HRV- 39.
  The inoculum is diluted, as appropriate, in lactated Ringer's solution and delivered via the following procedure: 0.5 ml per nostril is administered by pipette while the subject tilts their head back.
  Interventions: Biological: GMP-grade HRV-39; Procedure: Bronchoalveolar Lavage; Drug: Methacholine Inhalation Challenge; Procedure: Nasal Lavage; Procedure: Nasal Scrapings; Procedure: Bronchial Brushings; Procedure: Lung Mucosal Biopsy; Procedure: Allergen Skin Prick Testing; Procedure: Venipuncture; Procedure: Bronchoscopy; Procedure: Spirometry
- Healthy Non-Asthmatic Control Group (Active Comparator): Healthy volunteers. Subjects will be inoculated with a total dose of 1000 TCID50 of HRV- 39.
  The inoculum is diluted, as appropriate, in lactated Ringer's solution and delivered via the following procedure: 0.5 ml per nostril is administered by pipette while the subject tilts their head back.
  Interventions: Biological: GMP-grade HRV-39; Procedure: Bronchoalveolar Lavage; Drug: Methacholine Inhalation Challenge; Procedure: Nasal Lavage; Procedure: Nasal Scrapings; Procedure: Bronchial Brushings; Procedure: Lung Mucosal Biopsy; Procedure: Allergen Skin Prick Testing; Procedure: Venipuncture; Procedure: Bronchoscopy; Procedure: Spirometry

INTERVENTIONS:
Biological: GMP-grade HRV-39 — Experimental rhinovirus infection: an FDA approved, GMP-grade HRV-39 stock (gift from Dr. Ronald B. Turner, University of Virginia), which has now been approved by Health Canada for human experimental use, will be used in this study.
  Other Names: human rhinovirus; common cold
Procedure: Bronchoalveolar Lavage
Drug: Methacholine Inhalation Challenge — The purpose of this test is to determine if lung airways narrow by more than 20%, which confirms an asthma diagnosis.
Procedure: Nasal Lavage
Procedure: Nasal Scrapings — This process uses a rhinoprobe to gently scrape the mucosal lining of the nose
Procedure: Bronchial Brushings
Procedure: Lung Mucosal Biopsy
Procedure: Allergen Skin Prick Testing — For the purposes of this study, allergy skin testing will be done with the following aero-allergens: cat epidermis, dog epidermis, horse, grass mix, tree mix, weed mix, ragweed and house dust mite, along with a histamine positive control and a buffer & glycerol negative control.
Procedure: Venipuncture — Peripheral blood for assessment of neutralizing antibodies to HRV-39
  Other Names: Blood draw
Procedure: Bronchoscopy — A small flexible tube the size of a pencil, with a video-camera built into the tip (called a bronchoscope), will be inserted through the nose or mouth and down into the lungs.
Procedure: Spirometry

SUMMARY:
In this study, the following subjects will be exposed to human rhinovirus (HRV):

* those with classification of mild-moderate asthma
* healthy control subjects.

The investigators will study the kinetics of HRV-induced inflammatory and remodeling responses in a well characterized group of asthmatic subjects and compare these outcomes to those in a healthy, non-asthmatic control group.

DETAILED DESCRIPTION:
Although changes in the lungs, known as remodeling, are a feature of asthma, the causes and mechanisms involved in the process have not yet been found. Recently, it has been established that remodeling can be observed in children prior to a formal diagnosis of asthma. Clinical studies indicate that HRV, "common cold" infections, are a common cause of recurrent respiratory illnesses in childhood, and children with HRV-associated wheezing episodes have an increased risk of developing asthma. This led to the hypothesis that HRV infections may play a central role in the start of the airway remodeling leading to asthma.

The goal of this study is to determine if alterations in relevant airway remodeling growth factors differ between healthy controls and asthmatic subjects, pre- and post-HRV infection. These growth factors will be assessed in bronchoalveolar lavage (BAL) fluid and endobronchial biopsy tissues and correlated with viral levels in both nasal lavage and BAL fluid.

ELIGIBILITY:
Inclusion Criteria:

Asthmatics:

* Male or female volunteers with intermittent or persistent mild to moderate allergic asthma, as defined by GINA guidelines 39.
* Between ≥18 and ≤ 50 years of age.
* Objective evidence of variable airflow limitation (≥12% and at least 200mL post-bronchodilator reversibility from baseline), or airway hyperresponsiveness (PC20 methacholine <16mg/ml) at the screening visit or within past 24 months.
* Pre-bronchodilator spirometry at baseline; FEV1 ≥70% of predicted; FEV1/VC ≥50%.
* Atopic, as evidenced by positive skin prick tests to ≥1 common aero-allergen, where positive is defined by a wheal of ≥2 mm compared to the negative control.
* Not be exposed to sensitizing seasonal allergens for at least 4 weeks before the study. Chronic exposure to perennial allergens will be permitted.
* Asthma symptoms controlled by either inhaled β22-agonists alone, or by low or moderate dose ICS (≤800mcg of budesonide or equivalent per day), administered either as monotherapy or in a fixed-dose combination with a long-acting β22-agonist (LABA). The doses of these maintenance medications should have remained stable for the 4 weeks prior to the study screening phase (Visit 2).
* Stable asthma symptoms, with no history of asthma exacerbation requiring short burst prednisone treatment within the 3 months prior to study entry.
* Be a non-smoker, as defined as no smoking in past 12 months, and have a lifetime ≤ 10 pack-year smoking history.
* In good general health (other than asthma) without clinically significant medical history of other co-morbidities, and a BMI of ≤ 30 kg/m2.
* Have no history of any life threatening episode of asthma, as judged by the study physician; this may include, but not be limited to, prior ICU admission or intubation.
* Subjects, or their partners, must be using a reliable form of contraception continuously from 4 weeks prior, to 4 weeks post participation.

Non-Asthmatics:

* Male or female volunteers, ≥18 and ≤ 50 years of age, in good general health, without a clinically significant medical history and a BMI of ≤ 30 kg/m2.
* Non-asthmatic, as defined by history and normal spirometry (FEV1 ≥80% and FEV1/FVC ≥75% of predicted value).
* Normal airway responsiveness (PC20 methacholine ≥16 mg/ml).
* Non-atopic, as determined by skin prick tests to common aero-allergens, where positive test defined as a wheal of ≥ 2 mm compared to the negative control.
* Be a non-smoker for ≥1 year, and have a lifetime ≤ 10 pack-year smoking history of smoking.
* Subjects, or their partners, must be using a reliable form of contraception continuously from 4 weeks prior, to 4 weeks post participation.
* All potentially eligible study subjects must be willing to participate in study, and be able to provide written consent prior to starting the study. The study protocol and consent form will be approved by the Calgary Conjoint Health Research Ethics Board.

Exclusion Criteria:

* Presence of neutralizing antibodies to HRV-39 at the screening visit to a titer of ≥ 1:2.
* Have symptoms of an active viral respiratory tract infection (cold symptoms), corroborated by a score of 3 or higher on the Jackson cold symptom questionnaire, during the screening phase (Visit 3).
* Current pregnancy or positive urine pregnancy test at screening or during the study.
* Use of any of the following medications in preceding 4 weeks prior to study entry and during the study: : oral and topical antihistamines, leukotriene receptor antagonists, inhaled anticholinergics, non-steroidal anti-inflammatory drugs (NSAIDS), antibiotics and anti-viral medications, over the counter 'cold' and influenza remedies, including decongestants, and oral anticoagulants.
* Use of prednisone within the last 3 months.
* Current acute or chronic illness (including infection) or recent recovery (within 4 weeks) from acute illness which could, in the opinion of the study physician, alter inflammatory responses (e.g., influenza, cold or other respiratory infection, etc.). • Autoimmune disease or immunodeficiency, or any household contacts who are known to be immune deficient.
* Known allergy to lidocaine.
* Any other significant concomitant medical issue, or findings on physical examination or laboratory testing that, in the opinion of the study physician, may pose additional risks from participation in the study (including undergoing bronchoscopy), or which may impact the quality or interpretation of the data obtained from the study.
* Clinically significant pre-bronchoscopy safety assessment laboratory tests (CBC, INR, electrolytes and creatinine), as well as a positive urine pregnancy test on all female subjects of child-bearing age, will be done at visit 2 (day -26) and visit 5 (Day 0) prior to bronchoscopy on Day -7 and Day 4.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Bronchial Alveolar Lavage (BAL) Fluid Protein Levels | Day -7 and Day 4
  The primary endpoint will be the protein levels in BAL fluid at Day 4 (post-infection) minus the value at Day -7 (pre-infection) for each of MMP-9, VEGF amphiregulin and activin A.

SECONDARY OUTCOMES:
Quantitative Changes in Gene Expression Between Groups | Day -7 and Day 4
  Quantitative changes in gene expression between groups in BAL fluid, bronchial brushings, nasal scrapings and mucosal biopsies, for selected airway remodeling mediator genes, including MMP-9, amphiregulin, VEGF and activin A.
Changes in symptom scores, viral titers, spirometry, airway responsiveness (PC20 methacholine) and FeNO levels. | Day -7 and Day 4
Quantification of inflammatory cells in the lower airways, assessed in BAL fluid and bronchial biopsies. | Day -7 and Day 4
Correlation of gene expression and protein levels of selected mediators with viral titer, symptom scores and numbers of inflammatory cells in the upper and lower airways. | Day -7 and Day 4

CONTACTS AND LOCATIONS:
Overall Officials: David Proud, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada